CLINICAL TRIAL: NCT01071733
Title: Fracture Evaluated in Emergency Room by Ultra Sound
Acronym: FREEUS
Status: Withdrawn | Type: Observational
Why Stopped: study was never initiated due to logistic causes
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: FREEUS
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2012-09

CONDITIONS: Fracture; Ultrasonography
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- ultrasound wrist
- ultrasound finger
- ultrasound ankle

SUMMARY:
The purpose of this study is to compare fracture diagnostic, conventional x-ray versus ultrasound.

DETAILED DESCRIPTION:
to compare fracture diagnostic, conventional x-ray versus ultrasound in an emergency room department.

ELIGIBILITY:
Inclusion Criteria:

* Recent trauma to the wrist, ankle or fingers
* clinical exam by ER staff and x-ray indication.
* informed concent

Exclusion Criteria:

* open fracture
* wounds
* unstable fractures requiring cast immobilisation before x-ray
* multi traumatised patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients in emergency room
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2013-09 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mogens P Jensen, phd, md, Study Director — Dep. of Reumatology, Aarhus University Hospital, Denmark
Locations (1):
- Aarhus University Hospital Emergency Dep., Aarhus, Denmark